CLINICAL TRIAL: NCT07092189
Title: Anxiety Related to Colposcopy and the Impact of Pre-colposcopy Intervention by a Clinical Nurse
Brief Title: Colposcopy Anxiety and the Role of Pre-procedure Nursing Intervention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Josianne Pare, Principal investigator, Doctor and Associate Professor at the Department of Obstetrics and Gynecology, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-5032
Record Dates: First submitted 2025-07-19; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual- No pre-procedure counseling about colposcopy (Sham Comparator): Call from the clinical nurse to schedule the appointment without counseling
  Interventions: Other: Treatment as usual: regular call to schedule the appointment without pre-procedure conseilling
- Pre-colposcopy counseling from a clinical nurse (Experimental): In the intervention group, the clinical nurse conducted a structured pre-colposcopy counseling session covering the following topics: verification of the patient's understanding of the reason for the colposcopy referral, explanation of the cervical cytology result, the procedure of the colposcopy, expectations regarding pain, the role of HPV in the development of precancerous and cancerous cervical lesions, counseling on HPV vaccination, and smoking cessation."
  Interventions: Other: Pre-colposcopy counseling by a clinical nurse

INTERVENTIONS:
Other: Pre-colposcopy counseling by a clinical nurse — In the intervention group, the clinical nurse conducted a structured pre-colposcopy counseling session covering the following topics: verification of the patient's understanding of the reason for the colposcopy referral, explanation of the cervical cytology result, the procedure of the colposcopy, expectations regarding pain, the role of HPV in the development of precancerous and cancerous cervical lesions, counseling on HPV vaccination, and smoking cessation."
  Arms: Pre-colposcopy counseling from a clinical nurse
Other: Treatment as usual: regular call to schedule the appointment without pre-procedure conseilling — In the control group, patients simply received a phone call to notify them of their appointment and, upon arrival, were given an information sheet about colposcopy. No pre-colposcopy discussion was conducted.
  Arms: Treatment as usual- No pre-procedure counseling about colposcopy

SUMMARY:
Colposcopy is essential for the diagnosis and prevention of cervical cancer. However, receiving screening results and being informed of the need to undergo a colposcopic examination are significant sources of anxiety for patients. This randomized controlled study aims to evaluate the impact of an intervention by a clinical nurse prior to a first colposcopy on patients' situational anxiety. Secondary objectives include patient satisfaction, perceived pain during the examination, and the exploration of sociodemographic factors related to anxiety.

ELIGIBILITY:
Inclusion Criteria:

* People with a cervix
* 21-65 years old
* Speaking French
* Abnormal pap smears warranting a colposcopy

Exclusion Criteria:

* Refusal to participate
* Inability to provide consent.
* Having previously undergone a colposcopy.
* Being pregnant
* Having a reason for consultation other than an abnormal cytology result (such as VIN, VAIN, suspected cancer, vulvar dermatological issues, etc.).

Max Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Pre-procedure situational anxiety | On the day of the colposcopy procedure
  The pre-procedure situational anxiety is measured on the day of the colposcopy using the State Trait Anxiety Inventory (STAI). The STAI is a validated 20 item self report assessment device which includes separate measures of state and trait anxiety. The minimum value is 20 and the maximum value is 80. Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Pain level perceived during the colposcopy procedure measured by a visual analog scale (VAS scale) | Immediately after the colposcopy procedure
  We measured the pain level perceived during the colposcopy procedure using a visual analog scale ranging from 0 to 10. Highest scores indicated higher level of pain perceived during the procedure.
Patient's satisfaction level | Immediately after the colposcopy procedure
  Patient satisfaction levels were assessed using the standardized Patient's Experience and Attitude Colposcopy Eindhoven Questionnaire (PEACE-q). It is a validated 8-item user-friendly self-rating tool with with questions on: level of being informed, preoccupation, level of stress and level of ease created during consultation. The 8 items are rated on a 4-point Likert scale (final scores ranging from 8 to 32). Higher scores indicate a more positive experience of the colposcopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Josianne Paré, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CIUSS Estrie CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No